CLINICAL TRIAL: NCT05280678
Title: Evidence-based Selection of Orthodontic Miniscrews, Increasing Their Success Rate in the Mandibular Buccal Shelf: A Randomized, Prospective Clinical Trial
Brief Title: Success Rate of the Miniscrews in the Mandibular Buccal Shelf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Michał Sarul, Associate Professor, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 293/2007
Record Dates: First submitted 2022-01-10; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Class III Malocclusion
Keywords: miniscrew; orthodontics; skeletal anchorage
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: 200 Absoanchor® miniscrews (Dentos, South Korea) in two sizes: SH2018-10 (length 10 mm, ø 18-20 mm) and SH1514-08 (length 8 mm, ø 14-15 mm) were inserted in the mandibular buccal shelf of 100 Caucasians aged 20-50 years, diagnosed with Class III malocclusion that required en-masse distalization of the mandibular dentition. We designed our project as a split-mouth study, therefore each patient received both SH2018-10 and SH1514-08 miniscrews. The same orthodontist (M.S.) inserted the screws near the muco-gingival junction, following one surgical protocol. Miniscrews were loaded with orthodontic force (NiTi coil springs) of approximately 200 g, two weeks after the surgery. On the same visit patients were surveyed upon pain incidence lasting longer than 48 hours. Then TISAD stability and soft tissue condition were closely examined at each appointment. Miniscrews were considered long-term stable if they served as an anchorage until completion of distalization of the mandibular teeth.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SH2018-10 miniscrew side (Experimental): We designed our project as a split-mouth study, therefore each patient received both SH2018-10 and SH1514-08 miniscrews, randomly assigned to either left or right side. To do so, our nurse divided both miniscrew types into two halves and assigned symbols appropriate for blinding the intervention. Thus, two combinations of miniscrew sets aroused: 1. SH1514-08R and SH2018-10L or 2. SH1514-08L and SH2018-10R, which were placed separately in opaque packages marked consecutively from "1" to "100" and stored on the tray with dividers. One hundred cards, labeled accordingly, were placed in an envelope, from which the nurse blindly pulled the card just before the miniscrew insertion, this way assigning the set number to every patient. Thus both: the placement side and the screw size were random for clinician.
  Interventions: Procedure: Orthodontic miniscrew insertion in the mandibular buccal shelf
- SH1514-08 miniscrew side (Experimental): We designed our project as a split-mouth study, therefore each patient received both SH2018-10 and SH1514-08 miniscrews, randomly assigned to either left or right side. To do so, our nurse divided both miniscrew types into two halves and assigned symbols appropriate for blinding the intervention. Thus, two combinations of miniscrew sets aroused: 1. SH1514-08R and SH2018-10L or 2. SH1514-08L and SH2018-10R, which were placed separately in opaque packages marked consecutively from "1" to "100" and stored on the tray with dividers. One hundred cards, labeled accordingly, were placed in an envelope, from which the nurse blindly pulled the card just before the miniscrew insertion, this way assigning the set number to every patient. Thus both: the placement side and the screw size were random for clinician.
  Interventions: Procedure: Orthodontic miniscrew insertion in the mandibular buccal shelf

INTERVENTIONS:
Procedure: Orthodontic miniscrew insertion in the mandibular buccal shelf — Each patient received miniscrews in both sizes. The same orthodontist (M.S.) performed all the insertion procedures. Miniscrews were always placed in the mandibular buccal shelf, laterally to the first and second molar interproximal area, with angulation 30 degree to the bone surface, meaning that miniscrew angulation should be approximately the same as the axial inclination of the adjacent molar. Miniscrews were loaded with orthodontic force 2 weeks after the surgery. The investigated factors were:
  * long-term success rate of the miniscrews in the buccal shelf of the mandible (miniscrews were considered long-term stable if they served as an anchorage until completion of mandibular distalization, at least 9 months);
  * peri-implantitis development (enlargement of the gingiva and/or redness and/or tendency to bleed);
  * the patient's report of pain lasting longer than 48 hours after miniscrew insertion.

SUMMARY:
Stability of the orthodontic miniscrews placed in the mandible is still considered to bare higher risk of failure compared to other intraoral locations. The aim of our study was to determine the influence of the miniscrew size on their long-term stability, occurrence of oral mucosa inflammation and pain lasting over 48 hours after implantation.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy Caucasians
* mild Class III maloclussion that required an absolute anchorage for en-masse distalization in the mandible
* hypodivergent or normal angle between the maxillary and mandibular planes
* excellent oral hygiene

Exclusion Criteria:

* Hyperdivergent angle between the maxillary and mandibular planes
* unfavorable anatomical conditions - e.g. presence of a strong frenulum potentially irritating the miniscrew head during chewing and/or facial movement

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Assessing the stability of miniscrews | The first evaluation was performed 2 weeks after miniscrew insertion and then every 4-6 weeks (at follow-up visits) throughout the duration of distalization (up to 2 years).
  The mobility of the miniscrews was checked clinically with cotton tweezers at each visit. Miniscrews that could not sustain orthodontic force and required replacement because of mobility were considered failures.
Assessing the presence of peri-implantitis | The first evaluation was performed 2 weeks after miniscrew insertion and then every 4-6 weeks (at follow-up visits) throughout the duration of distalization (up to 2 years).
  Hypertrophy of the gingiva and/or redness and/or tendency to bleed was noted as the inflammation presence.
Assessing the presence of pain lasting longer than 48 hours after implantation. | two weeks
  Two weeks after the miniscrew implantation patients were surveyed upon pain incidence lasting longer than 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Michał Sarul, Principal Investigator — Wroclaw Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarul M, Lis J, Park HS, Rumin K. Evidence-based selection of orthodontic miniscrews, increasing their success rate in the mandibular buccal shelf. A randomized, prospective clinical trial. BMC Oral Health. 2022 Sep 20;22(1):414. doi: 10.1186/s12903-022-02460-3. PMID 36127718